CLINICAL TRIAL: NCT00778804
Title: Preventing Heart Disease in Underserved Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Geisinger Clinic (Other); Insight Telehealth Systems (Industry); Pennsylvania Department of Health (Other Government)
Responsible Party: Catherine Becker, Pennsylvania Department of Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4159
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Hypertension; Diabetes Mellitus; Hyperlipidemia
Keywords: CVD risk; self monitoring; Internet; telemedicine
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hyperlipidemias | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telemedicine (Experimental): Web-based monitoring in addition to usual clincial care with quarterly visits
  Interventions: Behavioral: telemedicine
- Control (No Intervention): Ususal care with quarterly visits

INTERVENTIONS:
Behavioral: telemedicine — Weekly transmission of health status (weight, activity, BP etc.) via the Internet with feeedback and reinforcement
  Arms: telemedicine

SUMMARY:
The study will evaluate the impact of an internet based telemedicine system on cardiovascular risk profile of underserved patient populations. It is our hypothesis that a treatment plan and frequent communication via an internet based Telemedicine system will improve the cardiovascular risk profile of underserved patient populations at increased risk for cardiovascular disease. Our primary endpoint is a reduction over one year in the 10-year CVD risk score (ATP III risk model).

DETAILED DESCRIPTION:
The Insight Telehealth system (ITSMyHealthfile) is a disease-managment interactive health care delivery system. Patients access the system through a special Web site using a password. The system prompts the patient to enter their weight, blood pressure and heart rate and there is a text box available for unstructed comments.

Patients will be randomized to either the telemedicine group or usual care group (controls). Individuals in the telemedicine group will be asked to transmit their health status weekly. Both groups will be followed for one year with quarterly visits.

Patients of either sex, of any ethnic background or race, between 22 and 85years of age, who have a 10% or greater 10-year risk of CVD based on the Framingham risk score, and risk factors that if properly treated would reduced the risk by 5% or greater will be eligible for the study.

Additional criteria

* literate
* telephone access
* ablility to utilize the Internet and telemedicine system (after training) Primary Outcome Reduction in Framingham risk index

ELIGIBILITY:
Inclusion Criteria:

* Framingham risk score equal to or greater than 10%
* literacy
* 22 -85 years of age
* access to phone

  * ability to use Internet and system following training

Exclusion Criteria:

* Class 3 and 4 heart failure
* ESRD
* stroke with residual disability or dementia
* unable to read or write

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2004-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Framingham 10-year risk index | 1 year

SECONDARY OUTCOMES:
Blood pressure, cholesterol, 6 minute walk test, glucose and A1c, CVD knowledge and risk perception | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Alfred A Bove, MD, PhD, Principal Investigator — Temple University
Locations (3):
- United States (3):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Temple University Hosptial, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Homko CJ, Deeb LC, Rohrbacher K, Mulla W, Mastrogiannis D, Gaughan J, Santamore WP, Bove AA. Impact of a telemedicine system with automated reminders on outcomes in women with gestational diabetes mellitus. Diabetes Technol Ther. 2012 Jul;14(7):624-9. doi: 10.1089/dia.2012.0010. Epub 2012 Apr 18. PMID 22512287
- [Derived] Bove AA, Santamore WP, Homko C, Kashem A, Cross R, McConnell TR, Shirk G, Menapace F. Reducing cardiovascular disease risk in medically underserved urban and rural communities. Am Heart J. 2011 Feb;161(2):351-9. doi: 10.1016/j.ahj.2010.11.008. PMID 21315219
- [Derived] McConnell TR, Santamore WP, Larson SL, Homko CJ, Kashem M, Cross RC, Bove AA. Rural and urban characteristics impact cardiovascular risk reduction. J Cardiopulm Rehabil Prev. 2010 Sep-Oct;30(5):299-308. doi: 10.1097/HCR.0b013e3181d6fb82. PMID 20436354